CLINICAL TRIAL: NCT04396873
Title: Phase 1 Study: PET Imaging of Cyclooxygenases in Neurodegenerative Brain Disease
Brief Title: PET Imaging of Cyclooxygenases in Neurodegenerative Brain Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200082; 20-M-0082
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-26

CONDITIONS: Parkinson's Disease; Dementia; Alzheimer's Disease; ALS; Mild Cognitive Impairment
Keywords: PET Imaging; PD; Inflammation; Dementia; Cyclooxygenase-2; ALS; MCI
MeSH Terms: conditions — Parkinson Disease; Dementia; Alzheimer Disease; Cognitive Dysfunction; Inflammation | interventions — (11C)-MC1; 11C-PS13; 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Only one arm (Other): All subjects receive the same tests
  Interventions: Drug: 11C-MC1; Drug: 11C-PS13; Drug: 18f-florbetaben

INTERVENTIONS:
Drug: 11C-MC1 — Injected IV followed by PET scanning
Drug: 11C-PS13 — Injected IV followed by PET scanning
Drug: 18f-florbetaben — Injected IV followed by PET scanning

SUMMARY:
Background:

About 5 million adults in the U.S. have Alzheimer s disease or another adult-onset neurodegenerative disorder. Many studies have found that inflammation in the brain contributes to these diseases. Researchers want to find a better way to measure this inflammation.

Objective:

To learn whether COX-1 and/or COX-2 is elevated in the brains of individuals with neurodegenerative brain disease compared to healthy volunteers.

Eligibility:

Adults age 18 years and older in good general health who have an adult-onset neurodegenerative dementia, such as AD, FTD, corticobasal syndrome, Huntington s disease, or MCI, ALS and healthy adult volunteers enrolled in protocols 01-M-0254 or 17-M-0181.

Design:

Participants will be screened with medical history, physical exam with vital signs, and lab tests. They will have a neuropsychological testing. Their heart function will be measured.

Participants will have a magnetic resonance imaging (MRI) scan. The MRI scanner is a metal tube surrounded by a strong magnetic field. Participants will lie on a table that slides in and out of the tube. The machine makes noise. Participants will get earplugs.

Participants will have 2 PET scans. They will be injected with the study drugs through an intravenous catheter placed in an arm vein. The PET scanner is shaped like a doughnut. Participants will lie on a bed that slides in and out of the scanner. A plastic mask will be molded to their head to keep them from moving. A thin plastic tube will be put into an artery at the wrist or elbow crease area. This will be used to draw blood during the scan.

Participants will have 2-5 study visits. Participation lasts 1 week to 4 months, depending on scheduling.

DETAILED DESCRIPTION:
Study Description:

This pilot/exploratory study will examine whether cyclooxygenase 1 (COX-1) and COX-2 are elevated in the brain of individuals with neurodegenerative brain disease compared to healthy volunteers.

Objectives:

Primary Objective: To determine whether COX-1 and/or COX-2 is elevated in the brains of individuals with neurodegenerative brain disease compared to healthy volunteers.

Secondary Objective:

1) To determine retest variability and reliability for each radioligand. 2) To evaluate the specific binding of [11C]PS13 to COX-1 in healthy subjects through blocking study using Ketoprofen, a COX-1 inhibitor

Endpoints:

Primary Endpoint: Measurement of COX-1 and COX-2 density in brain after PET scans with [11C]PS13 and [11C]MC1, respectively.

Secondary endpoint: 1) To measure whole-brain distribution volume (VT) of COX-1 and COX-2 in a retest setting; 2) To correlate VT with the presence of amyloid in Alzheimer s disease (AD) patients, mild cognitive impairment (MCI) patients and healthy volunteers (HV); 3) To calculate the specific binding of [11C]PS13 with a Lassen plot

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients: In order to be eligible to participate in this study, patients must meet all of the following criteria:

1. Aged 18 or older.
2. Be able (or have their Legally Authorized Representative (LAR) be able) to understand the study and be willing to sign a written informed consent document.
3. Have been diagnosed by a neurologist or psychiatrist with MCI, ALS, PD, or an adult onset neurodegenerative dementia, such as AD (including amyloid negative subjects), FTD, corticobasal syndrome, or Huntington s disease.
4. Be in good general health as evidenced by medical history and physical examination.
5. Have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
6. Agree to adhere to the lifestyle considerations.

Healthy volunteers: In order to be eligible to participate in this study, healthy volunteer subjects must meet all of the following criteria:

1. Aged 18 or older.
2. Female participants of childbearing potential must be using a medically acceptable means of contraception
3. Able provide informed consent.
4. Be in good general health, as evidenced by medical history and physical examination, and have no cognitive impairment.
5. Be enrolled in 01-M-0254, The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17-M-0181, Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies
6. Have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
7. Agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Both patients and healthy volunteers who meet any of the following criteria will be excluded from participation in this study:

1. Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen). Any lab value that is two-times the upper limit or even lower values in the investigator s judgment. Creatinine level >1.3 mg/dL
2. Subjects should not have taken Non-Steroidal Anti-Inflammatory Drugs (NSAID) for two weeks prior to the PET scan. Aspirin, corticosteroids (with the exception of skin products), or immunosuppressants (e.g., methotrexate) must not have been taken in the prior month.
3. Contraindications to ketoprofen, such as hypersensitivity to ketoprofen or history of upper or lower gastrointestinal bleeding.
4. Have other major neurological or medical diseases that may cause cognitive dysfunction, such as structural brain diseases, metabolic diseases, paraneoplastic syndromes, infectious diseases, or other significant neurological abnormalities.
5. Have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
6. Are unable to travel to the NIH.
7. Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
8. Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the patient and/or caregiver during the screening visit.
9. Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function of daily life.
10. Participants should not be under treatment with Aduhelm, nor should they have been treated in the past.
11. Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye).
12. Pregnancy
13. HIV infection
14. Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2029-04-11 (Estimated); Study Completion 2030-10-03 (Estimated)

PRIMARY OUTCOMES:
Measure the concentration of radioligands | 1-2 days
  Density of COX-1 and COX-2 in brain

SECONDARY OUTCOMES:
Measure the retest variability and reliability of the radioligans | 1-2 days
  Density of COX-1 and COX-2 in brain

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
results will be shared
Supporting Information: Study Protocol
Time Frame: 18 months after closure of protocol to Clincialtrials.gov
Access Criteria: BTRIS

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-M-0082.html